CLINICAL TRIAL: NCT03905109
Title: Phase 2b/3, Randomized, Double Blind, Placebo Controlled Induction Phase Followed by a Maintenance Phase to Evaluate the Efficacy & Safety of ABX464 in Patients With Moderate to Severe Active Crohn's Disease & to Determine the Optimal Dose
Brief Title: Phase 2b/3 Study of ABX464 in Moderate to Severe Active Crohn's Disease Patients
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Study design revised and to be found under new NCT06456593 ABX464-202
Sponsor: Abivax S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ABX464-201
Record Dates: First submitted 2019-04-03; First posted 2019-04-05 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Crohn Disease
Keywords: Inflammatory Bowel Disorders; ABX464
MeSH Terms: conditions — Crohn Disease | interventions — ABX464

STUDY DESIGN:
Intervention Model Description: Double-blind, placebo-controlled, randomized study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-Blind Treatment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ABX464 dose A (Experimental): Dose A QD
  Interventions: Drug: ABX464
- ABX464 Dose B (Experimental): Dose B QD
  Interventions: Drug: ABX464
- Placebo (Placebo Comparator): Matching dose
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ABX464 — ABX464 is a new anti-inflammatory drug. In the treatment arm, patients will receive dose A or Dose B of ABX464 orally once daily for 52 weeks.
  Arms: ABX464 Dose B; ABX464 dose A
Drug: Placebo — In the placebo group, patients will receive dose A or B ABX464-matching-placebo orally once daily for 52 weeks.
  Arms: Placebo

SUMMARY:
This is a multicenter, randomized, placebo controlled study to evaluate the efficacy and safety of ABX464, administered once daily (QD), in inducing clinical remission and endoscopic response in patients with moderate to severe active Crohn's disease (CD) who have inadequate response, loss of response, or intolerance to prior corticosteroid and/or immunosuppressant treatment and/or biologics. This study consists of a 28 day Screening Period, a 52 week Treatment Period; including a 12 week double blinded (Cohort 1) or open label (Cohort 2) Induction Phase and a 40 week double blinded (responders) or open label (nonresponders) Maintenance Phase; and a 4 week Follow up Period, which will consist of an End of Study (EOS) visit

DETAILED DESCRIPTION:
This is a multicenter, randomized, placebo controlled study to evaluate the efficacy and safety of ABX464, administered once daily (QD), in inducing clinical remission and endoscopic response in patients with moderate to severe active Crohn's disease (CD) who have inadequate response, loss of response, or intolerance to prior corticosteroid and/or immunosuppressant treatment and/or biologics. This study consists of a 28 day Screening Period, a 52 week Treatment Period; including a 12 week double blinded (Cohort 1) or open label (Cohort 2) Induction Phase and a 40 week double blinded (responders) or open label (nonresponders) Maintenance Phase; and a 4 week Follow up Period, which will consist of an End of Study (EOS) visit

Patient eligibility will be determined during a 4 week (28 days) Screening Period. Entry criteria will be based on confirmation of active moderate to severe ileal, ileocolic, or colonic CD. Approximately 930 patients will participate in this study (ABX464 Dose A N = 380, ABX464 Dose B N = 380, placebo N = 170).

On Day 0, eligible patients will be randomized into 2 cohorts:

* Cohort 1: Double blinded Induction Phase according to a 1:1:1 ratio into 3 treatment groups as follows:

  * ABX464 - Dose A QD: 170 patients
  * ABX464 - Dose B QD: 170 patients
  * Matching Placebo: 170 patients
* Cohort 2: Open-label Induction Phase according to a 1:1 ratio into 2 treatment groups as follows:

  * ABX464 - Dose A QD: 210 patients

At the end of the 12-week Induction Phase, all patients will be evaluated for the co-primary endpoints, namely induction of clinical remission and endoscopic improvement in addition to the secondary and exploratory endpoints. All patients will also be evaluated for treatment response. The determination of whether patients will be considered treatment responders versus nonresponders, responders being defined as patients with a reduction from baseline in Crohn's Disease Activity Index (CDAI) of ≥ 70 points.

Patients will be allocated to the different maintenance treatment regimens according to the following rules:

* Patients who received ABX464 in the Induction Phase (coming from Cohort 1 and 2) and who were responders at Week 12 will be randomized 1:1:1 to receive either ABX464 Dose A QD, ABX464 Dose B QD, or placebo in a double-blinded manner, for an additional 40 weeks. Stratification factors used for re-randomization in the Maintenance Phase are previous failure to biologics and current corticosteroid treatment use.
* Patients who received ABX464 or placebo in the Induction Phase (coming from Cohort 1 and 2) but who were not responders at Week 12 will be allocated to open label ABX464 Dose A QD. They will be evaluated 12 weeks later, and they will continue only if they have achieved clinical response at that timepoint.
* Patients who received placebo (coming from Cohort 1) in the Induction Phase and who were responders at Week 12 will be allocated to receive placebo as part of their double blinded maintenance treatment.

At Week 24, nonresponders who received open label ABX464 Dose A QD in the Maintenance Phase will be assessed for treatment response. If patients have not achieved treatment response at Week 24, patients should discontinue study drug. All patients, including those who have had treatment response in Week 12, can be discontinued due to disease worsening.

Patients will also be evaluated for safety and efficacy throughout the Induction and Maintenance Phases. From Day 0 onwards, all eligible patients will be followed at the investigational site on Week 1, Week 2, Week 4, Week 8, Week 12, and every 4 weeks until Week 52. Ileocolonoscopy will be performed in accordance with the Schedule of Activities.

ELIGIBILITY:
Inclusion Criteria:

* Men or women age 18-75 years;
* Patients must have a documented diagnosis (endoscopic with histology) of CD for ≥ 3 months before screening;
* Patients must have active moderate to severe ileal, ileocolic, or colonic CD at baseline as defined by 220 ≤ CDAI > 450,
* Patients must have a SES-CD score > 6 (≥4 if isolated ileal disease) at screening, assessed by ileocolonoscopy and confirmed by a central reading.
* Patients must be willing and able to undergo endoscopy during screening after all other inclusion criteria have been met and at the end of Week 16.
* Patients must have had either a documented inadequate response, no response, a loss of response, or an intolerance (defined as the occurrence of at least one Adverse Reaction leading to treatment discontinuation) to either amino-salicylates, immunosuppressant treatment (i.e., azathioprine, 6-mercaptopurine, methotrexate, biologics (i.e. tumor necrosis factor inhibitors, vedolizumab, ustekinumab), and/or corticosteroid treatment.
* Patients should be able and willing to comply with study visits and procedures as per protocol;
* Patients should understand, sign and date the written voluntary informed consent form at the screening visit prior to any protocol-specific procedures being performed;
* Patients should be affiliated to a social security regimen (for French sites only);
* Females and males receiving the study treatment and their partners must agree to use a highly effective contraceptive method during the study and for 3 months after end of study or early termination.

Exclusion Criteria:

* Patients with indeterminate colitis, microscopic colitis, ischemic colitis, infectious colitis, radiation colitis or clinical/histologic findings suggestive of ulcerative colitis;
* Patients with colonic dysplasia or neoplasia or adenomatous colonic polyp;
* Patients with presence of fistulae;
* Patients with current symptomatic diverticulitis or diverticulosis;
* Patients with obstructive colonic stricture/stenosis, past medical history of colonic resection, a history of bowel surgery within 6 months before screening, or who are likely to require surgery for CD during the treatment period;
* Patients with past medical history of clinically significant short bowel syndrome;
* Patients requiring parenteral nutrition;
* Patients with past medical history of bowel surgery resulting in an existing or current stoma;
* Patients with active infections at screening such as infected abdominal abscess, Clostridium difficile (stool antigen and toxin required), cytomegalovirus, tuberculous colitis and recent infectious hospitalization;
* Acute, chronic or history of clinically relevant pulmonary, cardiovascular, hepatic, pancreatic or renal functional abnormality, encephalopathy, neuropathy or unstable central nervous system pathology such as seizure disorder, angina or cardiac arrhythmias, or any other clinically significant medical problems as determined by physical examination and/or laboratory screening tests and/or medical history;
* Acute, chronic or history of immunodeficiency or autoimmune disease;
* History of malignancy excluding patients considered cure (5 years disease free survivors);
* Active malignancy that may require chemotherapy or radiation therapy;
* Serious illness requiring systemic treatment and/or hospitalization within 3 Weeks prior to baseline;
* Pregnant or breast-feeding woman;
* Illicit drug or alcohol abuse or dependence;
* Use of any investigational or non-registered product within 3 months or within 5 half-lives preceding baseline, whichever is longer;
* Any condition, which in the opinion of the investigator, could compromise the patient's safety or adherence to the study protocol.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-09-19 (Estimated); Primary Completion 2022-09-19 (Estimated); Study Completion 2022-09-19 (Estimated)

PRIMARY OUTCOMES:
The co-primary objectives of the study are to determine the efficacy of ABX464 in inducing clinical remission and endoscopic improvement after 12 weeks of study treatment in patients with moderate to severe active CD who have inadequate response, loss of | from baseline, at Week 12
  Percentage of patients in clinical remission at Week 12, defined as CDAI of ≤ 150
Co-primary objectives of the study are to determine the efficacy of ABX464 in inducing clinical remission and endoscopic improvement after 12 weeks of study treatment in patients with moderate to severe active CD who have inadequate response, loss of | from baseline, at Week 12
  Percentage of patients with endoscopic improvement at Week 12, defined as a decrease from baseline of ≥ 50% in the global SES-CD (SES CD 50)

SECONDARY OUTCOMES:
To evaluate the safety of ABX464 | from baseline, at week 12
  * Number and rate of all adverse events, causally related adverse events, all Serious Adverse Events (SAEs), and causally-related SAEs classified by severity
  * Incidence of treatment-emergent SAEs
  * Incidence of adverse events leading to investigational medicinal product discontinuation
  * The number of clinically-significant laboratory abnormalities
To evaluate the effect of ABX464 as measured by Patient-Reported-Outcome-based remission (PRO) at Week 12 | from baseline, at week 12
  Number and rates of patients with the following:
  PRO-based remission at Week 12, defined as abdominal pain ≤ 1 and liquid/soft Stool Frequence (SF) score of ≤ 3, averaged over the 7 days prior to visit
To evaluate the effect of ABX464 on C reactive protein (CRP) and fecal calprotectin levels | from baseline, at week 12
  Change from Week 0 to Week 12 in CRP and fecal calprotectin levels
To evaluate the effect of ABX464 on patients' quality of life | from baseline to week 12
  The scores and changes from Week 0 to Week 12 in Inflammatory Bowel Disease Questionnaire (IBDQ)
To evaluate the effect of ABX464 on micro RNA (miR) 124 expression in whole blood and in tissue | from baseline to week 12
  Change from Week 0 to Week 12 in microRNA-124 levels in total blood (PAXgene®) and in tissue (RNA later)
To assess the pharmacokinetics of ABX464 and ABX464-N-Glu | from baseline, at week 12
  Serum concentration of ABX464 and its main metabolite ABX464-N-Glu levels
To evaluate the effect of ABX464 as measured by endoscopic remission at Week 12 | from baseline, at week 12
  Number and rates of patients with the following:
  Endoscopic remission at Week 12 defined as SES CD ≤ 4 with at least a 2 point reduction from baseline
To evaluate the effect of ABX464 as measured by clinical response at Week 12 | from baseline, at week 12
  Number and rates of patients with the following:
  Clinical response at Week 12, defined as a reduction from baseline in CDAI of ≥ 100 points

CONTACTS AND LOCATIONS:
Overall Officials: Paul GINESTE, PharmD, Study Director — Abivax S.A.
Locations (1):
- University Hospitals Leuven - campus Gasthuisberg, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: Undecided